CLINICAL TRIAL: NCT07123896
Title: Arrhythmia Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025136
Record Dates: First submitted 2025-07-29; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Catheter Ablation; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment
  Interventions: Device: Normal treatment with catheter ablation or medicine; Drug: Drug Treatment

INTERVENTIONS:
Device: Normal treatment with catheter ablation or medicine — Routine clinical care with catheter ablation and/or medicine; real-world clinical cases
Drug: Drug Treatment — Routine clinical care with medicine; real-world clinical cases

SUMMARY:
The goal of this prospective, observational registry study is to evaluate the long-term effectiveness, safety, and impact of different kinds of treatment on the quality of life across diverse arrhythmia subtypes and patient populations in hospitalized adults with cardiac arrhythmias (including atrial fibrillation, atrial flutter, supraventricular tachycardia, and ventricular arrhythmias) undergoing routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for any type of arrhythmia

Exclusion Criteria:

* Patients currently participating in interventional clinical trials that may confound data collection or outcome assessment in this study.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for various types of arrhythmia
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-08-24 (Estimated); Primary Completion 2030-07-24 (Estimated); Study Completion 2030-07-24 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 1 year
  Recurrence of the arrhythmia after treatment
All-cause death | 1 year
  Death due to any reason

SECONDARY OUTCOMES:
Arrhythmia recurrence | 5 year
  Recurrence of the arrhythmia after treatment
All-cause death | 5 year
  Death due to any reason
Cardiovascular death | 1 year
  Death due to cardiovascular disease
Cardiovascular death | 5 year
  Death due to cardiovascular disease
Heart failure | 1 year
  Heart failure due to cardiovascular disease
Heart failure | 5 year
  Heart failure due to cardiovascular disease
Cardiovascular hospitalization | 1 year
  Hospitalization due to cardiovascular disease
Cardiovascular hospitalization | 5 year
  Hospitalization due to cardiovascular disease

CONTACTS AND LOCATIONS:
Locations (1):
- Deyong Long, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided